CLINICAL TRIAL: NCT06763770
Title: Digital Self-Management and Peer Mentoring Intervention to Improve the Transition From Pediatric to Adult Health Care for Childhood Cancer Survivors
Brief Title: Digital Self-Management and Peer Mentoring Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Southern California (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Katie Devine, PhD, MPH, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2023000838; R01CA282147 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Cancer Survivor; Survivorship; Cancer
Keywords: Pediatric cancer survivors; Self-management; Young adults; Childhood cancer survivors; Transition; Peer mentor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Managing Your Health (MYH) (Experimental): The Managing Your Health app + Peer Mentoring Intervention
  Interventions: Behavioral: Managing Your Health (MYH)
- Usual Care + Educational Control (Active Comparator): The Usual Care + Educational Control
  Interventions: Behavioral: The Usual Care + Educational Control

INTERVENTIONS:
Behavioral: Managing Your Health (MYH) — The Managing Your Health intervention consists of six weekly videoconference calls with a peer mentor and five self-management educational modules within a mobile application. The first call is to get to know each other, share survivorship stories, identify self-management strengths and weaknesses, and select goals for participation in the intervention. The remaining five weekly calls cover a self-management topic each week, including understanding your survivorship care plan, navigating the healthcare system and insurance, managing the emotional aspects of survivorship, negotiating family and significant other involvement in care, and engaging in healthy lifestyle behaviors.
  Arms: Managing Your Health (MYH)
Behavioral: The Usual Care + Educational Control — The Usual Care + Educational Control group will receive weekly emails with links to the Health Links developed by the Children's Oncology Group for use in survivorship care. Access to these Health Links reflects the current state of clinical care available to survivors. These Health Links were developed as patient education materials to cover relevant self-management and survivorship care topics. The weekly messages will align with the content of the modules from Managing Your Health to provide similar information, including Introduction to Long-Term Follow-Up (Module 1), Finding and Paying for Healthcare (Module 2), Emotional Issues (Modules 3 and 4), Educational Issues, Diet and Physical Activity, Skin Health, Reducing the Risk of Second Cancers, and Male/Female Health Issues (Module 5).
  Arms: Usual Care + Educational Control

SUMMARY:
This study tests how helpful a digital self-management and peer mentoring program is to young adult survivors of childhood cancer to improve their ability to manage their survivorship care as they transition from pediatric to adult-oriented follow-up care. Survivors require lifelong "risk-based" follow-up care based on the treatment they received to identify and treat late health effects. The transition from pediatric to adult follow-up care is a critical period when many survivors are lost to follow-up. Barriers to successful transition and engagement in care include poor knowledge of cancer history, low healthcare self-efficacy, poor self-management skills, low health literacy, and access issues such as financial hardship, insurance, and distance from cancer center. The "Managing Your Health" digital self-management and peer mentoring program aims to address these gaps and improve survivorship care self-management. Improvements in healthcare self-management are necessary to keep young adult survivors engaged in recommended health care, improve their quality of life, and promote optimal health.

DETAILED DESCRIPTION:
The purpose of the study is to determine the efficacy of the Managing Your Health intervention to improve self-management of survivorship care among young adult survivors of childhood cancer.

Aim 1: Evaluate the efficacy of the Managing Your Health intervention. Aim 2: Determine the mechanisms through which Managing Your Health influences outcomes.

Aim 3: Identify subgroups of participants for which treatment effects vary to inform future scale up.

Managing Your Health will be tested in a two-arm parallel randomized controlled trial (RCT) of the intervention versus usual care + educational control with 300 young adult survivors of childhood cancer currently aged 18-25 years. Participants will complete outcome measures at baseline, 3 months, and 12 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with any malignant childhood cancer between the ages 0-19 at least 5 years prior
2. Cancer treatment occurred at a pediatric center/facility
3. Current age 18-25
4. At least 2 years from treatment completion (typical time for transfer to long-term follow-up care)

Exclusion Criteria:

1. Any documented physical or self-reported cognitive delay that could prevent self-management of health care
2. Diagnoses of cancer not typically considered pediatric (I.e., melanoma, carcinoma of the breast, colorectum, lung, ovary, and testicle)
3. Unable to speak/read English

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Self-Management behaviors | Baseline, 3 months, 12 months
  The Self-Management Skills scale is a 15-item measure about a patient's active behaviors in managing their health. Response options were modified such that participants respond on a 5-point scale from 1 (not at all) to 5 (completely) regarding their agreement to each item. Example items include "I participate in making decisions about my health" and "I book my own doctor's appointments." A total mean score will be used, which could range from 0 to 5. Higher scores indicate better self-management behaviors.

SECONDARY OUTCOMES:
Adherence to guideline-concordant survivorship care | Baseline, 12 months
  Participants will report on cancer-specific and general medical appointments, surveillance tests, cancer screenings, and detection of new comorbidities using items from the Follow-Up Care Use Among Survivors (FOCUS) survey developed by NCI and items from surveys in the Childhood Cancer Survivor Study. Given the purposeful heterogeneity of our sample, we focus on the most common surveillance recommendations. We will report separately on receipt of cancer-related follow-up care (yes/no) and survivorship care plan (yes/no). For other tests, participants will be deemed adherent if they are up-to-date on recommended tests based on their health history. A summary score will be calculated for each participant by dividing the total number of recommendations completed by the total number of guideline-recommended tests. Thus, each participant will have a score that could range from 0 to 1, with 0 indicating no engagement in care and 1 indicating fully adherent to guideline concordant care.
Health-related Quality of Life | Baseline, 3 months, 12 months
  The Patient Reported Outcomes Measurement Information System (PROMIS) Global Health measure is a 10-item measure that assesses self-rated health, physical quality of life, mental quality of life, fatigue, pain, and participation in social activities and roles. The PROMIS measures have undergone extensive testing and are widely used. The Global Health measure yields a Physical Summary and Mental Health Summary scores, in addition to the total score. We will use the total score, which is standardized as a T-score with a mean of 50 and standard deviation of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Levonyan-Radloff, MS, Study Director — Rutgers Cancer Institute
Locations (2):
- United States (2):
  - University of South California, Los Angeles, California
  - Rutgers Cancer Institute, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will collect self-reported and medical-record data from 300 AYA survivors of childhood cancer. The final dataset will include self-reported demographic, psychosocial, and behavioral data from surveys as well as records of healthcare utilization. Documentation of the variables included in the dataset will be provided with the dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Even with removal of all identifiers, we believe there remains a very small possibility of identifying subjects with unusual characteristics. Therefore, we will make de-identified data available to qualified individuals within the scientific community for research purposes under a data-sharing agreement that specifies that data will only be used for research purposes, transfer of data will be done through secure methods, and investigators will commit to destroying copies of the data after analyses are completed.

REFERENCES:
- [Derived] Collins MKR, Levonyan-Radloff K, McLaughlin J, Masterson M, Devine KA. Designing an App to Facilitate Self-Management in Young Adult Survivors of Childhood Cancer: Development and Usability Study. JMIR Cancer. 2025 Dec 24;11:e77121. doi: 10.2196/77121. PMID 41442700